CLINICAL TRIAL: NCT00491309
Title: Exercise and Respiratory Therapy in Patients With Rheumatoid Arthritis / Collagenosis and Pulmonary Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Ekkehard Gruenig, Prof. Dr. med. Ekkehard Grünig, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Reha PH Rheumatic
Record Dates: First submitted 2007-06-25; First posted 2007-06-26 (Estimated); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Pulmonary Hypertension; Connective Tissue Disease
MeSH Terms: conditions — Hypertension, Pulmonary; Connective Tissue Diseases | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- exercise training group (Active Comparator): exercise and respiratory therapy with specific program for pulmonary hypertension (respiratory therapy, dumbbell training, ergometer training, mental training)
  Interventions: Behavioral: exercise training
- Control group without exercise training (No Intervention): continuation of sedentary lifestyle without advice for specific exercise training

INTERVENTIONS:
Behavioral: exercise training — exercise training with specific program (respiratory therapy, dumbbell training, ergometer training, mental training)
  Arms: exercise training group

SUMMARY:
In Patients with rheumatic disease exercise training is a well established element of therapy. In contrast patients with severe pulmonary hypertension are advised to avoid physical exertion and must not perform exercise training. This study aims to evaluate the effectivity and safety of a low-dose training program in patients with pulmonary hypertension and rheumatic disease.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent
2. Men and women 18 - 80 years
3. Diagnosed rheumatic disease: rheumatoid arthritis, Collagenosis (Systemic Lupus Erythematodes, Systemic Sclerosis, Sjögren-Syndrome, Sharp-Syndrome, Crest-Syndrome, Mixed connective tissue disease)
4. Symptomatic PAH (WHO- functional class II-IV) invasively diagnosed by right heart catheterisation

   * Mean pulmonary artery pressure (mPAP) > 25 mmHg
   * Pulmonary capillary wedge pressure (PCWP) > 15 mmHg
   * Pulmonary vascular resistance (PVR) at baseline >320 dyn.sec/cm5 patients under optimized medical treatment since at least 2 ½ months

Exclusion Criteria:

1. Other forms of PAH.
2. Pregnancy or lactation
3. Change in medication during the last 2 ½ months
4. Patients with signs of right heart decompensation
5. Severe impairment of walking
6. Unclear diagnosis
7. No invasive diagnosis of PH
8. Acute illness, infection, fever
9. Severe lung disease with FEV1 <50% and TLC< 70% below reference

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2011-07; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in the 6-minute walking distance | after 3 weeks and after 15 weeks compared to baseline.
Quality of life (SF-36) | baseline and 15 weeks

SECONDARY OUTCOMES:
change in inflammatory parameters (BKS, CRP, Leucocytes), change in inflammatory cytokines (TNF-α), change in parameters of the vascular endothelium (Endothelin, PDGF, VEGF), and endothelial progenitor cells | baseline and 15 weeks
Physical capacity in the cardiopulmonary exercise testing (Watt) | baseline, 3 weeks, 15 weeks
change of peak oxygen consumption and other parameters of cardiopulmonary exercise testing. | baseline, 3 weeks, 15 weeks
hemodynamic parameters: dimension and pump function of the right and the left ventricle. | baseline, 15 weeks
change in systolic pulmonary arterial pressure at rest and during exercise | baseline, 3 weeks, 15 weeks
  echocardiography
change of NTproBNP-value | baseline, 3 weeks, 15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ekkehard Gruenig, MD, Principal Investigator — Thoraxclinic at the University Hospital Heidelberg
Locations (1):
- Thoraxclinic at the University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Grunig E, Maier F, Ehlken N, Fischer C, Lichtblau M, Blank N, Fiehn C, Stockl F, Prange F, Staehler G, Reichenberger F, Tiede H, Halank M, Seyfarth HJ, Wagner S, Nagel C. Exercise training in pulmonary arterial hypertension associated with connective tissue diseases. Arthritis Res Ther. 2012 Jun 18;14(3):R148. doi: 10.1186/ar3883. PMID 22709477